CLINICAL TRIAL: NCT02748980
Title: Clinical Observation of Coronary Arterial Microcirculation Dysfunction in Diabetic Patients With Non- Obstructive Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhongwei, Attending doctor, Shaanxi Provincial People's Hospital
Other Study IDs: LHJJ20159029
Record Dates: First submitted 2016-04-17; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Complications of Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Complications; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Non- obstructive coronary artery disease, non- diabetic: Clinical evidences such as Holter, Treadmill exercise test and cardiac ECT support myocardial ischemia. CAG showed 20%-70% arterial stenosis. Patients are diagnosed without diabetes.
- Non- obstructive coronary artery disease, diabetic: Clinical evidences such as Holter, Treadmill exercise test and cardiac ECT support myocardial ischemia. CAG showed 20%-70% arterial stenosis. Patients are diagnosed with type 2 diabetes.

SUMMARY:
The purpose of this study is to investigate the prevalence and degree of coronary arterial microcirculaiton dysfunction of non- obstructive coronary artery disease in patients with type 2 diabetes. Furthermore, the risk factors of coronary arterial microcirulation would be screened and identified.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis non- obstructive coronary artery disease;
* Positive Treadmill exercise test;
* Positive Cardiac ECT test;
* Positive Holter test

Exclusion Criteria:

* Diagnosis of myocardial infarction;
* Diagnosis heart failure;
* Diagnosis of chronic kidney disease;
* Diagnosis of heart valvular disease;
* Diagnosis of malignant tumor;
* Positive heart transplant history;
* Pregnant and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The coronary microcirculation dysfunction is measured by index of microcirculatory resistance | 10 minutes after diagnosis is made by CAG

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial People's Hospital, Xi'an, Shaanxi, China